CLINICAL TRIAL: NCT03379883
Title: Combined Ultrasound Guided Genicular Nerve and Intra-articular Pulsed Radiofrequency Versus Intra-articular Platelet Rich Plasma Injection for Chronic Knee Osteoarthritis; A Comparative Study
Brief Title: Genicular Nerve and Intra-articular Radiofrequency Versus Platelet Rich Plasma Injection for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD/17.01.37
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Chronic Knee Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blind (investigator) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed radiofrequency (P-RF) (Placebo Comparator): Patients will receive both intra articular RF and genicular nerve RF ablation
  Interventions: Procedure: Pulsed radiofrequency (P-RF)
- Platelet rich plasma (PRP) (Experimental): Patients will receive intra-articular platelet rich plasma (PRP)
  Interventions: Procedure: Platelet rich plasma (PRP)

INTERVENTIONS:
Procedure: Pulsed radiofrequency (P-RF) — Intra articular RF
  Insertion of the RF cannula within the joint. The recommended parameters are a pulse width of 20 msec and a rate of 2 Hz at 42°C for 10min.
  Genicular nerve RF ablation.
  The RF probe will be placed. A 50 Hz-frequency sensorial stimulation will be applied with a threshold of < 0.6 V
  Arms: Pulsed radiofrequency (P-RF)
Procedure: Platelet rich plasma (PRP) — Under ultrasound guidance while the patients in a sitting position. In total, 3 to 8 mL of PRP will be injected via the inta-articular route
  Arms: Platelet rich plasma (PRP)

SUMMARY:
The social impact of degenerative diseases such as articular cartilage pathology and osteoarthritis (OA) is steadily increasing, because of the continued rise in the mean age of the active population. A variety of noninvasive solutions have been proposed for pain treatment, improvement in function and disability, and ultimately, modification of the course of severe cartilage lesions and OA, with variable success rates. Intra articular and genicular nerves radiofrequency (RF) is a minimally invasive technique that usually aims at the neuropathic pain. One important mechanism for the chronic pain mediated by OA is peripheral sensitization, which increases the transmission of pain signals. Through conduction block in pain-transmitting nerve fibers by thermal damage, RF could ease pain without destroying the antennal nerve. The role of growth factors (GFs) in chondral repair is now widely investigated in vitro and in vivo.

Platelet-rich plasma (PRP) is a simple, low cost, and minimally invasive method that allows one to obtain from the blood a natural concentrate of autologous GFs.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of intra articular Platelet Rich Plasma (PRP) injection versus combined ultrasound guided intra articular and genicular nerve pulsed radiofrequency on chronic knee pain in patients with knee osteoarthritis.

The regeneration capacity of cartilage is limited because of its isolation from systemic regulation and its lack of vessels and nerve supply. Osteoarthritis (OA) has a major impact on functioning and independence and ranks among the top 10 causes of disability worldwide

ELIGIBILITY:
Inclusion Criteria:

* Patients experienced unilateral lesion with a history of chronic (≥4 months)
* Pain or swelling of the knee and imaging findings (radiography or magnetic resonance imaging [MRI]) of degenerative changes of the joint
* Patients shall to be clinically unresponsive to conservative treatment modalities

Exclusion Criteria:

* Diabetes
* Rheumatic diseases
* Coagulopathies
* Severe cardiovascular diseases
* Infections
* Immunosuppression
* Patients receiving anticoagulants
* Use of non-steroidal anti-inflammatory drugs in the 5 days before blood donation
* Hemoglobin concentration less than 10 g/dl
* Platelet count less than 150,000/cubic mm.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | For 6 months after intervention
  The intensity of pain at rest will be measured with a 10-cm visual analogue scale (VAS-pain). (VAS) identifying 0 as no pain and 10 as worst imaginable pain.

SECONDARY OUTCOMES:
Knee function | For 6 months after intervention
  Subjective knee functionality will be evaluated using the Western Ontario and McMaster's Universities Osteoarthritis (WOMAC) Index.WOMAC Index assesses disability in three subscales, including pain, severity of physical function and joint stiffness. This scale consists of 24 items: five items for pain assessment, two items for assessment of the severity of joint stiffness and 17 items for assessment of physical function. The patient answers the questions and then receives a cumulative score in each of the 3 areas (pain, 0-20; stiffness, 0-8; physical function, 0-68). Higher scores are representative of greater pain and stiffness as well as worsened physical capability.
Patient satisfaction | For 6 months after intervention
  Patient satisfaction when it comes to perceived improvement in symptoms after the treatment will evaluated using the Patient Global Impression Scale of Improvement (PGI-I) where; Very much better = 1, Much better = 2, A little better= 3, No change =4, A little worse=5, Much worse=6, Very much worse =7,

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Sultan, MD, Principal Investigator — Professor of Anesthesia and Surgical Intensive Care; Doaa G Diab, MD, Study Chair — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Emergency Hospital, Intensive Care Unit, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided